CLINICAL TRIAL: NCT04541771
Title: The Role of Lactobacillus Reuteri (L. Reuteri) in Preventing Necrotizing Enterocolitis (NEC) in Pre-term Infants Less Than 34 Weeks of Gestation
Brief Title: The Role of Lactobacillus Reuteri in Preventing Necrotizing Enterocolitis (NEC) in Pre-term Infants
Acronym: NEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital and Institute of Child Health, Multan (Other Government)
Responsible Party: Principal Investigator, Dr Summera Tabasum, post-graduate resident, Children's Hospital and Institute of Child Health, Multan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CH&ICH
Record Dates: First submitted 2020-08-05; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Necrotizing Enterocolitis; Sepsis
Keywords: Necrotizing Enterocolitis,; lactobacillus reuteri ds 17938
MeSH Terms: conditions — Enterocolitis, Necrotizing; Sepsis

STUDY DESIGN:
Intervention Model Description: participants will be divided in two groups. one is control group and the other Interventional group. control group will receive the drug under study and control will be given placebo for the period of until they complete 35 weeks of gestation or discharged.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- drug group (Experimental): The trial group will receive their usual feeds plus daily probiotic (Lactobacillus Reuteri DSM 17938) addition 1 drop/kg/dose(. minimum of 20 million live Lactobacillus Reuteri are present in One drop) twice daily added in expressed breast milk/formula milk from the beginning of enteral feedings till the baby attain full feeds
  Interventions: Drug: Lactobacillus Reuteri DSM 17938
- control group (Placebo Comparator): this group is control group and will receive normal saline drops as 1 drop/kg/ dose mixed in enteral feed
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus Reuteri DSM 17938 — The trial group will receive their usual feeds plus daily probiotic addition 1 drop/kg/dose twice daily added in expressed breast milk/formula milk from the beginning of enteral feedings till the baby attain full feeds
  Arms: drug group
Drug: Placebo — expressed breast milk/formula milk plus normal saline drop from the beginning of enteral feedings till the baby attain full feeds
  Arms: control group

SUMMARY:
The purpose of this study is to compare the effectiveness of L. Reuteri with placebo in prevention of NEC in children, as according to my knowledge, there is limited work is done nationally and internationally. Probiotics are being used in our Children Hospital and the Institute of Child Health, Multan.

Route of administration of L. Reuteri will be oral or via nasogastric tube due to availability of oral form in Pakistan. The results of this study will be helpful to assess the beneficial effects of probiotics especially L. Reuteri in NEC in preterm. So, they can be recommended as preventive strategy to avoid NEC development and its complications based on its availability, effectivity and easy administration

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonate< 34 weeks and >28 weeks of gestation of both genders Hemodynamically stable

Exclusion Criteria:

* Preterm neonates >34 weeks gestational age < 28 weeks of gestation Cardiorespiratory illness Parental refusal

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
narcotizing enterocolitis | up to 35 weeks of gestation
  number of participants with the sign of feeding intolerance (such as the gastric aspirate in the amount that was more than half of previous feeding), or with abdominal distension measured by increase in abdominal girth from base line,Bell Staging Criteria according to clinical and radio-logical signs

SECONDARY OUTCOMES:
sepsis | At time of addmission and 15 days after intervention
  number of participants who developed sepsis proven by blood cultures before of after intervention

CONTACTS AND LOCATIONS:
Overall Officials: summera tabasum, Principal Investigator — CH&ICH